CLINICAL TRIAL: NCT07274839
Title: Digitalization Through the Use of Ren'Py-Based Interactive Learning Experiences in Physiotherapy and Rehabilitation Education: A Randomised, Controlled, Single-Blind Study
Brief Title: Interactive Ren'Py Learning in Physiotherapy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmet Koçyiğit (Other)
Responsible Party: Sponsor-Investigator, Ahmet Koçyiğit, Lecturer, Zonguldak Bulent Ecevit University
Organization: Zonguldak Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 03.07.2024/468499; https://osf.io/38ntm (Other: Open Science Framework)
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Student

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three groups-Conventional Education Group (CEG), Digital Education Group (DEG), or Conventional and Digital Education Group (CaDEG)-using a random sequence generated via random.org
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Education (Active Comparator): The course content was standardized using materials from the "CK4Stim-Clinical Key for Electrical Stimulation in Physiotherapy and Rehabilitation" project (CK4Stim, Access Date: October 2024). The CK4Stim project, supported by the European Union and involving multiple projects partners, aims to develop a common language for the use of electrical stimulation in physiotherapy and rehabilitation education in accordance with European standards.
  Interventions: Other: Conventional Instructional Material
- Digital Education (Experimental): A lesson package containing a story in an interactive visual novel format created using Ren'Py. This package was designed by the researchers to include the theoretical and practical contents of the medium frequency currents unit, again using the content of the CK4Stım project.
  Interventions: Other: Digital Instructional Material
- Conventional and Digital Education (Other): A group that received both educational models for comparison.
  Interventions: Other: Digital Instructional Material; Other: Conventional Instructional Material

INTERVENTIONS:
Other: Digital Instructional Material — A lesson package containing a story in an interactive visual novel format created using Ren'Py. This package was designed by the researchers to include the theoretical and practical contents of the medium frequency currents unit, again using the content of the CK4Stim project.
  Arms: Conventional and Digital Education; Digital Education
Other: Conventional Instructional Material — The course content was standardized using materials from the "CK4Stim-Clinical Key for Electrical Stimulation in Physiotherapy and Rehabilitation" project (CK4Stim, Access Date: October 2024). The CK4Stim project, supported by the European Union and involving multiple projects partners, aims to develop a common language for the use of electrical stimulation in physiotherapy and rehabilitation education in accordance with European standards.
  Arms: Conventional Education; Conventional and Digital Education

SUMMARY:
Advances in health professions education increasingly emphasize the use of digital technologies to enhance student engagement and support diverse learning needs. In physiotherapy training, particularly in technically complex subjects like electrotherapy, conventional instruction may fall short in fostering active learning and knowledge retention. Game-based platforms such as Ren'Py offer an opportunity to integrate interactive, scenario-based learning into the curriculum. This study aimed to assess the impact of Ren'Py-based digital materials on learning outcomes by comparing conventional, digital, and hybrid teaching models in an undergraduate electrotherapy course.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Cumulative GPA above 1.80
* Access to a device compatible with at least one of the following operating systems or platforms: Linux x86_64/Arm, Windows 7 or later, or Mac OS X 10.10 or later

Exclusion Criteria:

* History of course failure due to absenteeism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Theoretical Knowledge Examination Score | Measured at 1-week follow-up after completion of the educational intervention.
  A researcher-developed 20-item multiple-choice theoretical exam assessing students' knowledge of electrotherapy principles.
  Full Scale Name: Theoretical Knowledge Examination (20-item multiple-choice test) Score Range: 0 to 100 points Interpretation: Higher scores indicate better theoretical knowledge.
Practical Skills Examination Score | Measured at 1-week follow-up after completion of the educational intervention.
  A 16-item practical performance assessment evaluated by an independent three-member exam jury. Each item was rated as "Sufficient", "Partial", or "Insufficient", and final scores were calculated as the arithmetic mean of the three jury evaluations, scaled to a 0-100 range.
  Full Scale Name: Practical Skills Performance Assessment (16-item jury-rated evaluation) Score Range: 0 to 100 points Interpretation: Higher scores indicate better practical performance.

SECONDARY OUTCOMES:
Cognitive Load Rating Score | Measured at 1-week follow-up after completion of the educational intervention.
  Subjective cognitive load was assessed using the nine-point Cognitive Load Rating Scale developed by Paas and Van Merriënboer (1993). Participants rated the level of mental effort experienced during the learning activity on a nine-point Likert-type scale.
  Full Scale Name: Paas & Van Merriënboer Cognitive Load Rating Scale (9-point Likert scale) Score Range: 1 (Very Low) to 9 (Very High) Interpretation: Higher scores indicate greater perceived cognitive load.
Instructional Materials Motivation Scale Score | Measured at 1-week follow-up after completion of the educational intervention.
  Motivation toward the instructional materials was assessed using the 33-item Instructional Materials Motivation Scale (IMMS) developed by Keller. Participants rated each item on a five-point Likert scale evaluating attention, relevance, confidence, and satisfaction related to the instructional materials.
  Full Scale Name: Instructional Materials Motivation Scale (IMMS), 33-item Likert scale Score Range: 33 (minimum) to 165 (maximum) Interpretation: Higher scores indicate higher motivation toward the instructional materials.

OTHER OUTCOMES:
Attitude Toward the Physiotherapy Profession Score | Assessed at baseline (prior to the intervention) and again 1 week after completion of the intervention.
  Attitudes toward the physiotherapy profession were measured using the Attitude Toward the Physiotherapy Profession Scale developed by Turhan. The scale contains 35 items rated on a five-point Likert scale and assesses three dimensions: professional satisfaction, required professional competencies, and general concerns regarding the profession.
  Full Scale Name: Attitude Toward the Physiotherapy Profession Scale (35-item Likert scale) Score Range: 35 (minimum) to 175 (maximum) Interpretation: Higher scores indicate more positive attitudes toward the physiotherapy profession.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Facultu of Health Sciences, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data and software repositories will be shared on OSF.

REFERENCES:
- [Derived] Kocyigit A, Cavlak U. Digitalization through the use of Ren'Py-Based interactive learning experiences in physiotherapy and rehabilitation education: a randomised, controlled, single-blind study. BMC Med Educ. 2025 Dec 22. doi: 10.1186/s12909-025-08474-z. Online ahead of print. PMID 41430217